CLINICAL TRIAL: NCT02686359
Title: Research of a Biological Marker for Chronic Orofacial Pain: Dosage of Opiorphin in Patients With Burning Mouth Syndrome
Brief Title: Opiorphin Levels in Fluids of Burning Mouth Syndrome Patients (OPIODYN)
Acronym: OPIODYN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P081106
Record Dates: First submitted 2016-02-05; First posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Burning Mouth Syndrome
Keywords: physiology; pain; analgesia; saliva; opiorphin
MeSH Terms: conditions — Burning Mouth Syndrome; Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Burning Mouth Syndrome Patients (Experimental): saliva, blood and urinary samples
  Interventions: Biological: sample
- controls (Active Comparator): saliva, blood and urinary samples
  Interventions: Biological: sample

INTERVENTIONS:
Biological: sample

SUMMARY:
If epidemiological studies indicate relatively low prevalence reported in the general population, idiopathic burning mouth syndrome (BMS) is a common condition among certain groups of the population: 30% of menopausal women experience oral burning to varying degrees . Despite significant progress made in recent years, in understanding the physiopathogeny, treatment options remain limited and disappointing,resulting in an impairment of the quality of life. Given the chronic nature of idiopathic burning mouth syndrome, the need to identify the causes and effective treatment modalities for subjects suffering is essential.

DETAILED DESCRIPTION:
Idiopathic burning mouth syndrome (BMS) is a chronic orofacial pain condition in which the pain is felt as intense, located on the tongue and the oral mucosa with no known cause. The pain may last for years and present treatments are of little effect. BMS is primarily a feminine disease, affecting women during or following menopause, suggesting an etiopathogenic role of the sexual hormones potentiating a local salivary factor. An anxiodepressive component is often associated with the disease. Recently, a molecule named opiorphin has been identified in human saliva. In animals, this molecule has shown potent analgesic properties comparable to those of morphine. The hypothesis of the investigators is that this molecule is in lower quantity in the saliva of persons suffering BMS and that this decrease causes oral burning sensations.

The main objective of the study is to test the hypothesis of a decrease of opiorphin levels in the saliva of patients suffering from primary BMS compared to a group of control subjects. The main judgment criteria is the level of salivary opiorphin in ng/mL.

The proposed study is a multicentric, simple blinded case controlled study. The investigators will collect the data from 21 primary BMS patients and 21 control subjects matched in sex, age, and hormonal status (menopause). The alpha risk is 0.5% and the power of the study is 90%.

Criteria for inclusion : BMS patients will be suffering for more than 4 months from burning pain in the tongue or oral mucosa with no organic trouble detectable by anamnesis, clinical evaluation and biological testing.

The design of the study includes three sessions for all subject of both groups; the maximum duration of participation for a subject is 8 weeks and the total duration of the study is 24 months There are two investigation centers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Burning Mouth Syndrome
* Age between 18 and 80 years
* Sensation of pain in the oral mucosa, meeting the diagnostic criteria for BMS (Bergdahl and Anneroth, 1993, Scala 2003)
* Signature of informed consent

Healthy volunteers

* Age between 18 and 80 years
* Patient age (+/- 5 years), sex and hormonal status (menopause or not for women) matched with a Burning Mouth Syndrome patient
* Signature of informed consent

Exclusion Criteria:

* Dental or periodontal pain during the month before the visit
* General pathology likely to cause mouth pain (diabetes, lupus, shingles, gastric reflux, allergies ...)
* Chronic Orofacial pain other than Burning Mouth Syndrome
* Treatment with a molecule able to induce oral burning sensations (anti-VEGF, neuroleptics, IEC angiotensin II ...)
* Participation concomitantly in biomedical research
* No affiliation to a social protection system
* Taste disorder other than a dysgeusia linked to Burning Mouth Syndrome
* Inability to understand the information note and sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
opiorphin levels in saliva | Day 30

SECONDARY OUTCOMES:
opiorphin levels in blood | Day 30
urinary levels in urine | Day 30

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boucher Y, Braud A, Dufour E, Agbo-Godeau S, Baaroun V, Descroix V, Guinnepain MT, Ungeheuer MN, Ottone C, Rougeot C. Opiorphin levels in fluids of burning mouth syndrome patients: a case-control study. Clin Oral Investig. 2017 Sep;21(7):2157-2164. doi: 10.1007/s00784-016-1991-0. Epub 2016 Nov 10. PMID 27834029